CLINICAL TRIAL: NCT01174901
Title: Copeptin for Risk Stratification in Non-traumatic Headache in the Emergency Setting - The CoHead Study
Acronym: CoHead
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CoHead
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Head Pain
Keywords: cephalalgia; copeptins; biomarkers; headache; C-terminal provasopression; physiological stress response
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 7.5 ml of EDTA blood, 7.5 ml of serum, 4.3 ml of citrate blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Headache is a common symptom, and patients often seek medical attention at emergency departments due to headaches.

The aim of the CoHead Study is to find out if it is possible by measuring copeptin, a marker of stress in the blood, to find out which patients have simple headaches and which patients have dangerous headaches that are the symptom of an underlying disease and need further investigation and treatment.

Copeptin is a marker for physical stress and has been tested in patients with stroke, heart attack and pneumonia. In all these illnesses, the patients with the most serious forms had the highest levels of copeptin, while the ones with only mild presentation or no affection at all had the lowest levels of copeptin.

The investigators expect to show the same in patients with headaches.

DETAILED DESCRIPTION:
Background: In the emergency setting, non-traumatic headache (NTH) is in 80% a benign symptom, but serious causes have to be ruled out.

Copeptin, as a surrogate marker for antidiuretic hormone (ADH), is a marker for the individual stress level, even more subtle than cortisol. As a prognostic stress hormone it holds promise as a prognostic point of care tool in the risk stratification of different acute illnesses such as acute myocardial infarction, respiratory tract infections and cerebrovascular events, among others.

Objective: To evaluate copeptin as a marker for risk stratification in NTH. Design: Prospective multicenter observational cohort study with a derivation set and a validation set.

Location Setting: Emergency Department (ED) and Medical Policlinic (MUP; walk-in clinic) and Neurologic Clinic (NC) of the University Hospital of Basel. ED and NC of the Cantonal Hospital of Aarau.

Intervention: Patients presenting to the ED or the MUP or the NC with NTH are recruited during a 1-year-period. After informed consent is given by the patient, baseline data will be assessed including medical history, clinical items (i.e. neurological status, vital parameters, blood pressure, BMI) and routine laboratory items. Patients will be evaluated using a validated standardized diagnostic tool and questionnaire. CT scans and other diagnostics, such as lumbar puncture, MRI, etc., will be ordered upon request of the treating physician. All diagnostic procedures, results, diagnosis made by the treating physicians and initiated therapy will be recorded. Copeptin will be measured on admission by batch analysis by blinded laboratory staff upon completion of the study.

After 3 months, all patients will be followed-up by a structured telephone interview to assess the final diagnosis and outcome (i.e. MIDAS-Questionnaire). The final diagnosis will be made by two independent physicians according to ICHDII-criteria and verified by a board-certified neurologist, all blinded to copeptin levels. Thereby, primary and secondary headache entities will be classified according to ICHD.

Endpoints: The primary endpoint of this study is serious secondary NTH as opposed to benign, self-limiting NTH. Serious secondary NTH will be defined as a composite endpoint including different secondary NTH causes and entities as listed in the International Classification of Headache Disorders (ICHD)-II-Criteria.

The secondary endpoint will be clinical outcome of patients; thereby we will look at all-cause mortality within the 3-month follow-up period and at morbidity measured by the MIDAS-questionnaire.

Study hypothesis: We hypothesize that copeptin will serve as a point of care tool to discriminate benign headache from potentially serious secondary headaches (e.g. subarachnoidal hemorrhage (SAH) or cerebral aneurysm, intracranial bleeding (ICB), brain tumor, vasculitis, meningitis) which require prompt hospitalisation and intervention. Based on copeptin values measured in other acute diseases, we assume a critical range between 5 and 20 pmol/l. The lower copeptin cutoff point of ≤ 5 pmol/l will have a sensitivity of ≥ 97% for ruling out serious secondary headache, and the higher cutoff point of ≥ 20 pmol/l will have a specificity of 90% to confirm serious NTH.

Analysis: Based on data of two previous years, we aim to recruit 600 - 800 patients within one year at the sites of Basel and Aarau, respectively, of which 10-20% will present with serious secondary NTH. We will calculate 95% confidence intervals of sensitivity of copeptin of <10% and perform multivariable logistic regression analysis to assess the independent and additive utility of copeptin compared with other risk scores and outcome predictors. The first 50% of patients will be used as derivation set and the second 50% as the validation set, based on the timely inclusion of patients.

Significance: If copeptin as a biomarker safely rules out serious secondary causes of NTH, it will represent a tool for an optimized allocation of health care resources.

ELIGIBILITY:
Inclusion Criteria:

* headache at the time of screening
* Patients must be able to give informed consent

Exclusion Criteria:

* less than 18 years of age
* preceding (head) trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to emergency department or walk-in clinic
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Differentiation between serious secondary non-traumatic headache as opposed to benign, self-limiting non-traumatic headache by copeptin level measurement | At study entry, assessment of baseline characteristics, questionnaire, further investigations done by attending physician, and blood collection for copeptin measurement. telephone interview after 3 months.
  Assessment of the prognostic value of copeptin to predict the primary endpoint (serious secondary NTH).
  Non-traumatic headache (NTH) will be assessed and defined according to the ICHD-II-Criteria. Serious secondary NTH will be defined as a composite endpoint including different secondary NTH causes and entities as listed in the ICHD-II-Criteria.

SECONDARY OUTCOMES:
clinical outcome of patients | study entry and 3-month-interview
  * all-cause mortality within the 3-month follow-up period
  * morbidity measured by the MIDAS-questionnaire which is performed at study entry and at the 3-month-interview
Additive benefit on sensitivity if copeptin and a diagnostic algorithm are combined | study entry and 3-month-interview
  A validated, diagnostic algorithm consisting of four clinical scenarios (published by Grimaldi et al.) will be used by the study team upon entry into the study. We will evaluate the additive benefit of copeptin to this algorithm with means of multivariate logistic regression analysis and calculation of reclassification tables.
Comparison of copeptin with other potential biomarkers in non-traumatic headache | study entry and 3-month-interview
  We will compare the diagnostic and prognostic accuracy of copeptin with other potential biomarkers which have been reported to be of diagnostic value in migraine or cerebrovascular events, both being potential clinical scenarios of non-traumatic headache.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, PhD, Principal Investigator — Department of Endocrinology, University Hospital of Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Kantonsspital Aarau AG, Aarau, Canton of Aargau
  - University Hospital of Basel, Basel, Canton of Basel-City

REFERENCES:
- [Background] Katan M, Fluri F, Morgenthaler NG, Schuetz P, Zweifel C, Bingisser R, Muller K, Meckel S, Gass A, Kappos L, Steck AJ, Engelter ST, Muller B, Christ-Crain M. Copeptin: a novel, independent prognostic marker in patients with ischemic stroke. Ann Neurol. 2009 Dec;66(6):799-808. doi: 10.1002/ana.21783. PMID 20035506
- [Background] Katan M, Muller B, Christ-Crain M. Copeptin: a new and promising diagnostic and prognostic marker. Crit Care. 2008;12(2):117. doi: 10.1186/cc6799. Epub 2008 Mar 6. PMID 18355399
- [Background] Reichlin T, Hochholzer W, Stelzig C, Laule K, Freidank H, Morgenthaler NG, Bergmann A, Potocki M, Noveanu M, Breidthardt T, Christ A, Boldanova T, Merki R, Schaub N, Bingisser R, Christ M, Mueller C. Incremental value of copeptin for rapid rule out of acute myocardial infarction. J Am Coll Cardiol. 2009 Jun 30;54(1):60-8. doi: 10.1016/j.jacc.2009.01.076. PMID 19555842
- [Background] Friedman BW, Hochberg ML, Esses D, Grosberg B, Corbo J, Toosi B, Meyer RH, Bijur PE, Lipton RB, Gallagher EJ. Applying the International Classification of Headache Disorders to the emergency department: an assessment of reproducibility and the frequency with which a unique diagnosis can be assigned to every acute headache presentation. Ann Emerg Med. 2007 Apr;49(4):409-19, 419.e1-9. doi: 10.1016/j.annemergmed.2006.11.004. Epub 2007 Jan 8. PMID 17210203
- [Background] Grimaldi D, Cevoli S, Cortelli P. Headache in the emergency department. How to handle the problem? Neurol Sci. 2008 May;29 Suppl 1:S103-6. doi: 10.1007/s10072-008-0899-0. PMID 18545909
- [Derived] Blum CA, Winzeler B, Nigro N, Schuetz P, Biethahn S, Kahles T, Mueller C, Timper K, Haaf K, Tepperberg J, Amort M, Huber A, Bingisser R, Sandor PS, Nedeltchev K, Muller B, Katan M, Christ-Crain M. Copeptin for risk stratification in non-traumatic headache in the emergency setting: a prospective multicenter observational cohort study. J Headache Pain. 2017 Dec;18(1):21. doi: 10.1186/s10194-017-0733-2. Epub 2017 Feb 13. PMID 28197843